CLINICAL TRIAL: NCT06125236
Title: Registration of Acute Ischemic Stroke With Large and Medium-sized Vascular Occlusion in Southwest China(LMVOS)
Acronym: LMVOS
Status: Recruiting | Type: Observational
Sponsor: Zhengzhou Yuan (Other)
Responsible Party: Sponsor-Investigator, Zhengzhou Yuan, Deputy Director of Stroke Center, The Affiliated Hospital Of Southwest Medical University
Organization: The Affiliated Hospital Of Southwest Medical University (Other)
Other Study IDs: SWMU202309
Record Dates: First submitted 2023-11-06; First posted 2023-11-09 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Thrombosis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute ischemic stroke with large- or medium-vessel occlusion: Acute ischemic stroke patients with large- or medium-vessel occlusion including all treatments.
  Interventions: Other: Visit at D90

INTERVENTIONS:
Other: Visit at D90 — Visits at 90±7 days after stroke onset were conducted by trained and blinded investigators, with face-to-face, telephone call or Internet access.

SUMMARY:
This study is designed to observe the treatment options in real-world clinical practice as well as the safety and efficacy of different treatment strategies.

DETAILED DESCRIPTION:
LMVOS is a prospective, real-world registry lasting for 22 years. A total of 8000 patients with large- or medium-vessel occlusion will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

The clinical diagnosis is acute ischemic stroke with large- or medium- vessel occlusion (the criteria followed the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2018).

Informed consent from the patient or surrogate.

Exclusion Criteria:

No additional exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute ischemic stroke due to large- or medium-vessel occlusion will be enrolled and no additional exclusion criteria are set.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2023-11-09 (Actual); Primary Completion 2045-12-01 (Estimated); Study Completion 2046-05-01 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score | 90±7 days
  Ordinal distribution of mRS at 90±7 days; modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)

SECONDARY OUTCOMES:
Excellent functional outcome | 90±7 days
  Proportion of subjects with mRS 0-1 at 90±7 days.
Good functional outcome | 90±7 days
  Proportion of subjects with mRS 0-2 at 90±7 days.
mRS 0-3 | 90±7 days
  Proportion of subjects with mRS 0-3 at 90±7 days.
Change of National Institutes of Health Stroke Scale (NIHSS) | 24 hours
  Change of National Institutes of Health Stroke Scale (NIHSS, a scale between 0 and 42 on which higher scores indicate more severe neurologic deficits) from baseline to 24 hours.
Change of National Institutes of Health Stroke Scale (NIHSS) | 7 days
  Change of National Institutes of Health Stroke Scale (NIHSS, a scale between 0 and 42 on which higher scores indicate more severe neurologic deficits) from baseline to 7 days.
Symptom-to-thrombolysis time (STT) | 24 hours
  Time from onset of symptoms to thrombolytic therapy.
Door-to-Needle Time | 24 hours
  Time from the arrival of stroke patient in emergency to initiation of thrombolysis therapy.
Door-to-Puncture Time (DPT) | 24 hours
  ime from the arrival of stroke patient in emergency to groin puncture.
Onset-to-recanalization time | 24 hours
  Time from symptom onset to the beginning of recanalization (recanalization defined as expanded TICI scale≥2b).
Door-to-Recanalization Time (DRT) | 24 hours
  Time from the arrival of stroke patient in emergency to the beginning of recanalization (recanalization defined as expanded TICI scale≥2b).
Puncture-to-recanalization time | 24 hours
  Time from groin puncture to recanalization (recanalization defined as expanded TICI scale≥2b).

OTHER OUTCOMES:
Incidence of clinically significant intracranial hemorrhage | 36 hours
  Incidence of sICH (Heidelberg criteria) measured at 36 hours
Incidence of any intracranial hemorrhage | 36 hours
  Incidence of any intracranial hemorrhage (Heidelberg criteria) measured at 36 hours
All-cause mortality | 90±7 days
  All-cause mortality at 90±7 days
Complications related to intravenous thrombolysis | up to 7 days
  Complications related to intravenous thrombolysis during hospitalization
Complications related to endovascular treatment | up to 7 days
  Complications related to intravenous thrombolysis during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Zhengzhou Yuan, MD, Study Chair — Department of Neurology, Affiliated Hospital of Southwest Medical University, LuZhou, China.
Locations (1):
- Affiliated Hospital of Southwest Medical University, Luzhou, China

IPD SHARING:
Plan to Share IPD: No